CLINICAL TRIAL: NCT01489098
Title: Effect of the Level of Dietary Protein on Infant Growth and Body Composition in the First Year of Life - Three and Five Year Growth and Body Composition Follow-up
Brief Title: Effect of the Level of Dietary Protein on Body Composition
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 06.29.INF Addendum
Record Dates: First submitted 2011-12-02; First posted 2011-12-09 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2014-10

CONDITIONS: Growth Acceleration
Keywords: Body composition; Protein Metabolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breast Fed reference group: 3 and 5 year olds from the above group
- Infant formula - protein level 1: 3 ad 5 year olds from the above group
- Infant formula - protein level 2: 3 and 5 year olds from the above group

SUMMARY:
The purpose of this study is to determine if toddlers and children who were fed breast milk or infant formulas at different levels of protein between 3 and 12 months of age have differences in growth and body composition at 3 and 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in infant formula controlled protein study
* Body composition data from 6 month of age available
* Consent obtained from legal representative
* Within age parameters specified in protocol around the 3 and 5 year age points

Exclusion Criteria:

* Unable to endure testing procedures upon evaluation of the Investigator
* Outside the age range of the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Toddlers and Children who have previously participated in an infant formula trial where various levels of protein were provided and who are now at the age of 3 and 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Mean weight gain | 3 years
Mean weight gain | 5 years

SECONDARY OUTCOMES:
Body composition | 3 years
Body composition | 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Samuel J Fomon Infant Nutrition Unit Department of Pediatrics, University of Iowa, Iowa City, Iowa
  - Department of Pediatrics, University of Oklahoma Health Sciences, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831